CLINICAL TRIAL: NCT04585724
Title: Evaluation of Radiosurgery With Concurrent Cyclin-Dependent Kinase 4/6 Inhibitors in the Treatment of Brain Metastases
Brief Title: Stereotactic Radiosurgery With Abemaciclib, Ribociclib, or Palbociclib in Treating Patients With Hormone Receptor Positive Breast Cancer With Brain Metastases
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed due to low (0) accrual
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jim Zhong, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000194; NCI-2019-02251 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD4615-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Anatomic Stage IV Breast Cancer American Joint Committee on Cancer (AJCC) v8; Metastatic Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — abemaciclib; palbociclib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment (abemaciclib) (Experimental): Beginning within 2 weeks prior to stereotactic radiosurgery, patients receive abemaciclib PO BID. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Other: Quality-of-Life Assessment
- Treatment (palbociclib) (Experimental): Beginning within 2 weeks prior to stereotactic radiosurgery, patients receive palbociclib PO QD on days 1-21. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Palbociclib; Other: Quality-of-Life Assessment
- Treatment (ribociclib) (Experimental): Beginning within 2 weeks prior to stereotactic radiosurgery, patients receive ribociclib PO QD on days 1-21. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Drug: Ribociclib

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
  Arms: Treatment (abemaciclib)
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
  Arms: Treatment (palbociclib)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011
  Arms: Treatment (ribociclib)

SUMMARY:
This phase I trial studies the side effects of stereotactic radiosurgery with abemaciclib, ribociclib, or palbociclib in treating patients with hormone receptor positive breast cancer that has spread to the brain (brain metasteses). Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to normal tissue. Abemaciclib, ribociclib, and palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving abemaciclib, ribociclib, or palbociclib concurrently with stereotactic radiosurgery may reduce the side effects and/or increase the response to each of the therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Prospectively evaluate safety and toxicity of the combination of radiosurgery (SRS) and concurrent CDK 4/6 inhibitors (CDKi) for hormone receptor positive (HR+) breast cancer patients.

SECONDARY OBJECTIVES:

I. Evaluate late toxicity (after 3 months) following SRS and concurrent CDKi. II. Evaluate local control efficacy with combination therapy of SRS and concurrent CDKi.

III. Assess quality of life and neurologic functional outcomes following treatment using standardized questionnaire (Functional Assessment of Cancer Therapy-Brain [FACT-Br]).

IV. Analyze overall survival.

OUTLINE: Patients are assigned to 1 of 3 groups.

GROUP I: Beginning within 2 weeks prior to stereotactic radiosurgery, patients receive abemaciclib orally (PO) twice daily (BID). Treatment continues in the absence of disease progression or unacceptable toxicity.

GROUP II: Beginning within 2 weeks prior to stereotactic radiosurgery, patients receive ribociclib PO once daily (QD) on days 1-21. Treatment continues in the absence of disease progression or unacceptable toxicity.

GROUP III: Beginning within 2 weeks prior to stereotactic radiosurgery, patients receive palbociclib PO QD on days 1-21. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 4-6 weeks post stereotactic radiosurgery, and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of hormone receptor positive (estrogen receptor >= 1 percent or progesterone receptor >= 1 percent) with HER2 negative status, past treatment, or systemic disease status with current clinical diagnosis of up to 10 brain metastases based on contrast-enhanced magnetic resonance imaging (MRI) of the brain
* Plan to start or currently receiving an Food and Drug Administration (FDA)-approved CDK4/6 inhibitor (CDKi), which must be started no later than 2 weeks prior to planned radiosurgery with plan to continue CDKi following radiosurgery
* Up to 10 brain metastases =< 3 centimeters in greatest dimension, measured on radiation planning MRI
* Eastern Cooperative Oncology Group (ECOG)/Zubrod 0-1, or Karnofsky performance status 70-100
* Contrast-enhanced MRI brain within 4 weeks of radiosurgical intervention (radiation planning MRI)
* Patients must be able to sign informed consent prior to study entry, including assent to standard of care post-treatment surveillance contrast-enhanced magnetic resonance imaging of the brain
* Patients who are enrolled in the study, and who continue to be prescribed CDK4/6 inhibitor therapy and develop new brain metastases deemed treatable by radiosurgery, are specifically allowed to be re-treated while on study, and the new treated lesions will be separately counted by treatment category (1 to 3, 4 to 6, or 7 to 10 new treated lesions)
* Patients with prior treated brain metastases (radiosurgery, hypofractionated radiotherapy, or surgery) are eligible for the study regardless of prior history of asymptomatic or symptomatic radiation necrosis and may not be excluded from the study if that is the sole basis for exclusion

Exclusion Criteria:

* Patients with current or prior invasive malignancy unless disease free for minimum of 1 year
* Brain metastases > 3 cm
* Brain lesions causing midline shift or herniation > 1 cm
* Patients with unirradiated post-neurosurgical metastasectomy resection cavities, unless disease-free in the surgical bed for >= 6 months, are prohibited from pilot study enrollment
* No patients who require resection cavity radiation for treatment of a resected brain metastasis (i.e.: standard of care treatment) are eligible for enrollment
* Receipt of chemotherapeutic agents (other than CDK4/6 inhibitors or hormone receptor-related targeted agents) within 2 weeks of planned radiosurgery date
* Prior whole brain or craniospinal radiotherapy
* Fractionated radiation to unrelated central nervous system (CNS) tumor
* Concurrent malignant CNS tumor
* Recurrent or progressive brain metastasis necessitating surgical or medical intervention (i.e.: a non-radiotherapy intervention such as steroids)
* Recurrence or progressive brain metastasis from prior surgical resection necessitating surgical or medical intervention (i.e.: a non-radiotherapy intervention)
* Brain stem metastasis >= 1 cm
* Patients with scleroderma
* Severe acute co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization in the last 3 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization in the last 6 months or precluding study therapy due to inability to rest supine at the time of registration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3+ radiation therapy oncology central nervous system toxicity | At 3 months
  Rate and frequency of grade 3+ toxicity will be reported. A 95% exact confidence interval will be estimated using the Clopper-Pearson method.

SECONDARY OUTCOMES:
Symptomatic radiation necrosis (late toxicity) | At 6 and 12 months
  Will be defined as radiographic (typically on magnetic resonance imaging) changes consistent with radiation induced necrosis and the patient presenting with increased neurological symptoms. Rate and frequency of late toxicity will be reported, and a 95% exact confidence interval will be estimated. Symptomatic radiation necrosis similarly will be summarized. The rate of radiation necrosis will be compared with that of our institutional historical control.
Intracranial failure within treated lesion | Up to 1 year
  Will be defined by progressive lesion either biopsy-proven or with imaging interpretation concordance by both radiation oncologist and neuroradiologist on serial imaging. The cumulative incidence approach will be used to estimate the failure rates for intracranial failure of treated lesion and distant intracranial failures.
Distant intracranial failure | Up to 1 year
  New lesions will be defined by new contrast-enhancing brain lesions on magnetic resonance imaging. The cumulative incidence approach will be used to estimate the failure rates for intracranial failure of treated lesion and distant intracranial failures.
Overall survival | Up to 1 year
  The Kaplan-Meier method will be used to estimate the overall survival rates.
Quality of life (QoL) | Up to 1 year
  Will be assessed by Functional Assessment of Cancer Therapy-Brain (FACT-Br) at pre- and post-radiosurgery. Will be summarized using frequencies and percentages for categorical variables, and mean, standard deviation, median, and range for continuous variables. Paired tests such as paired t-tests and McNemar's tests will be considered for comparing QoL outcomes pre- versus post-radiosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jim Zhong, Principal Investigator — Emory University